CLINICAL TRIAL: NCT03110224
Title: Zimmer Knee Creations SCP® Observational Cohort Follow-Up Study
Brief Title: SCP® Observational Study of the Knee
Status: Terminated | Type: Observational
Why Stopped: Enrollment of 500 subjects was met and Sponsor decided to discontinue enrollment as of July 2018. Sponsor believes enrollment number will provide us with sufficient follow-up to submit a substantial manuscript with minimum of 2 year follow-up data.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: KC.CR.I.AM.16.3
Record Dates: First submitted 2017-03-28; First posted 2017-04-12 (Actual); Results first posted 2025-08-27 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2024-12

CONDITIONS: Bone Marrow Edema
Keywords: Subchondroplasty; Bone Marrow Lesion; Arthroscopy; Bone Substitute Material; AccuFill; Subchondral Bone Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Subchondroplasty Procedure with AccuFill — Injection of the commercially available flowable calcium phosphate (CaP) synthetic bone-void filler, AccuFill®, into subchondral bone defects in the knee(Subchondroplasty (SCP) Procedure).

SUMMARY:
Post Market clinical outcomes study to collect data on the short - and long-term outcomes for subjects who are undergoing or who have undergone the Subchondroplasty (SCP) Procedure in the knee in a standard clinical setting. Outcomes to be assessed include pain medication usage, pain, function, activity levels and patient satisfaction.

DETAILED DESCRIPTION:
This is a post-market, multi-center, patient outcomes centered study to evaluate the on-label use of AccuFill during the Subchondroplasty procedure. Enrolled subjects will sign an informed consent form, satisfy the inclusion/exclusion criteria and have at least one Bone Marrow Lesion (BML) in the knee. Demographics, medical history and medications will recorded at the time of enrollment. Surgical details including the SCP procedure, concomitant surgical procedures and intraoperative safety events will be recorded. Subjects will complete patient reported outcomes measures pre-operatively including the Visual Analog Scale (VAS) for knee pain, International Knee Documentation Committee Subject Knee (IKDC) Form and the Veterans Rand 12 (VR-12) Item Health Survey. These measures will also be administered post-operatively at 6 weeks, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years. Screening for adverse events and revision surgeries will occur throughout the study.

Target enrollment is 1000 subjects at up to 30 clinical sites. Subjects will complete the study at 5 years or will be withdrawn if the patient undergoes revision surgery of the Subchondroplasty site.

ELIGIBILITY:
Inclusion Criteria:

1. Surgeon considers patient appropriate for SCP procedure.
2. Patient has agreed to undergo the SCP procedure or has already undergone the procedure.
3. Subject is willing and able to sign a written consent form.
4. The subject has the mental capacity and the willingness to contribute follow-up outcome data.
5. Patient is willing and able to complete outcome forms in person or by phone, email or regular mail.

Exclusion Criteria:

1. Patient is not comfortable with speaking, reading, and understanding questions and providing responses in an available language for the PROs in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The SCP Observational Cohort Study will enroll either patients undergoing SCP or patients who have already had the SCP procedure for the treatment of BMLs where bone void filler is placed at the site of the BML (defect).
Sampling Method: Non-Probability Sample
Enrollment: 516 (Actual)
Dates: Start 2012-09-18 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Jaggard, Study Director — Zimmer Biomet
Locations (14):
- United States (14):
  - Denver-Vail Orthopedics, Parker, Colorado
  - Atlantis Orthopaedics, Palm Beach Gardens, Florida
  - Foundation for Orthopaedic Research and Education (FORE), Tampa, Florida
  - Southern Ortho, Johns Creek, Georgia
  - OrthoIndy, Indianapolis, Indiana
  - Cascio Sports Medicine, Lake Charles, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Orthopaedic Surgical Associates, North Chelmsford, Massachusetts
  - Beaumont Health System, Royal Oak, Michigan
  - Associated Orthopedists, Saint Clair Shores, Michigan
  - New York University School of Medicine, Huntington Station, New York
  - Ohio State University, Columbus, Ohio
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Jordan-Young Institute, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Subchondroplasty® (SCP®) Procedure — https://www.subchondroplasty.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 516 patients enrolled, 508 had data entered that could be used for analysis.
Groups:
- Subchondroplasty: Patients who were to undergo Subchondroplasty
Period: Overall Study
Arm/Group | Subchondroplasty
Started | 516
Completed | 133
Not Completed | 383
Not completed — Death | 3
Not completed — Lost to Follow-up | 132
Not completed — Physician Decision | 2
Not completed — Site Closed by Physician | 35
Not completed — Site Closed by Sponsor | 202
Not completed — Withdrawal by Subject | 9

BASELINE CHARACTERISTICS:
Groups:
- Baseline: Demographics of patients enrolled in the study.
Arm/Group | Baseline
Number analyzed (Participants) | 516
Age, Categorical [Count of Participants; unit: Participants] — Population: 2 patients did not have age entered at baseline
  Participants
    number analyzed (Participants) | 514
    <=18 years | 0
    Between 18 and 65 years | 299
    >=65 years | 215
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 2 patients did not have age entered at baseline.
  years
    Age: number analyzed (Participants) | 514
    Age | 56.77 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender not entered for 8 patients
  Participants
    number analyzed (Participants) | 508
    Female | 272
    Male | 236
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 516
BMI [Mean (Standard Deviation); unit: kg/m2] — Population: BMI could not be calculated for 12 patients due to missing weight, height, or both.
  kg/m2
    number analyzed (Participants) | 504
    (all) | 31.53 (6.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Visual Analog Scale (VAS) Pain Scale at 12 Months
Description: Change from baseline score of pain intensity at 12 months. To collect VAS, patients marked a slash on a 10 cm horizontal line, with 0 cm indicating "no pain" and 10 cm indicating "worst possible pain." The distance from the left end of the line to the patient's mark was measured by the administrator in centimeters. Lower numbers were representative of lower pain levels.
Time Frame: 12 months
Population: Visual Analog Scale was analyzed at baseline to 12 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Primary Outcome Measure: Visual Analog Scale measured at baseline and 12 months.
Arm/Group | Primary Outcome Measure
Number analyzed (Participants) | 250
score on a scale
  Baseline | 6.8 [6.6 to 7.0]
  12 Months | 3.6 [3.3 to 4.0]

2. Secondary Outcome: Occurences and Severity of Device and/or Procedure Related Adverse Events and Re-visions/Re-operations
Description: Summary and description of procedure and device related adverse events and surgical re-operations and relatedness to the bone substitute material and procedure
Time Frame: 5 years
Measure: Number; unit: Number of Events Reported
Groups:
- Secondary Outcome Measure: Summary and description of procedure and device related adverse events and surgical re-operations and relatedness to the bone substitute material and procedure
Arm/Group | Secondary Outcome Measure
Number analyzed (Participants) | 508
Number of Events Reported
  Events Related to SCP | 36
  Events Unrelated to SCP | 72
  Revisions | 72

ADVERSE EVENTS:
Time Frame: Surgery, 6 weeks, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
Groups:
- Adverse Events: Adverse Events reported during the study.
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 3/516
Serious Adverse Events (participants affected / at risk) | 83/516
Other Adverse Events (participants affected / at risk) | 17/516
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=516)
Chondrosis: Patella and Medial Femoral Condyle (Musculoskeletal and connective tissue disorders) | 1 (1)
Complex tear of medial meniscus of right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Extensive chondrosis medial femoral condyle and medial tibial plateau (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Increased grinding and retropatellar pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Infected right knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Known patellar chondrosis with recurrent effusions and pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 47 (49)
Osteoarthritis with fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Persistence of patellofemoral pain not responsive to conservative management. (Musculoskeletal and connective tissue disorders) | 1 (1)
Post-operative pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Femoral Popliteal DVT (Blood and lymphatic system disorders) | 1 (1)
Septic Knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Subchondral edema/stress fracture reaction medial femoral condyle and medial tibial plateau (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left knee draining sinus (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain secondary to pancreatic cancer stage 2 A (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone marrow lesion in femur (Musculoskeletal and connective tissue disorders) | 1 (1)
Cephalgia (General disorders) | 1 (1)
Complete tear of medial and lateral menisci (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Knee Pain (Musculoskeletal and connective tissue disorders) | 11 (11)
L4-5 Laminectomy w posterior fusion O-arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Laparoscopic sleeve gastrectomy w PEH repair for morbid obesity BMI 45.0-49.9 (Gastrointestinal disorders) | 1 (1)
Left shoulder scope w rotator cuff repair (Musculoskeletal and connective tissue disorders) | 1 (1)
Parapatellar increased synovium and scar (Musculoskeletal and connective tissue disorders) | 1 (1)
Persistently symptomatic chondral defect of patella (Musculoskeletal and connective tissue disorders) | 1 (1)
Persistently symptomatic patellar cartilage defect (Musculoskeletal and connective tissue disorders) | 1 (1)
Persistently symptomatic patellar chondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Right Eye Cataract (Eye disorders) | 1 (1)
Right Knee arthroscopy (non study knee) (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Total knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=516)
Acute Cholecystitis (Gastrointestinal disorders) | 1 (1)
Arthroscopic Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Difficulty with dorsiflexion of left foot. (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee draining sinus (Musculoskeletal and connective tissue disorders) | 1 (1)
Left knee stress fracture lateral femoral condyle and impending OCD lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Medial femoral condyle insufficiency fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Patient had signs of delirium postoperatively (General disorders) | 1 (1)
Right knee chondromalacia patella with right thigh muscle/tendon strain. (Musculoskeletal and connective tissue disorders) | 1 (1)
Stress fracture left foot (Musculoskeletal and connective tissue disorders) | 1 (1)
GI virus (Gastrointestinal disorders) | 1 (1)
Patient reported knee popping with pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Total knee arthroplasty (Musculoskeletal and connective tissue disorders) | 1 (1)
Unicompartment knee replacement (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Follow-up compliance: Fewer than half of enrolled participants completed follow-up at or beyond 2 years.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT03110224/Prot_SAP_001.pdf